CLINICAL TRIAL: NCT04865016
Title: Clinical Outcomes With a Low Add Multifocal and an Extended Depth of Focus Intraocular Lenses Both Implanted With Mini-monovision
Brief Title: Low Add Multifocal Versus Extended Depth of Focus Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2016.309
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Multifocal Intraocular Lenses; Extended Depth of Focus
Keywords: low add multifocal intraocular lens, MIOL, ZKB00, extended depth of focus, EDOF, ZXR00, mini-monovision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIOL Group (Active Comparator): 30 eyes of 15 cataract patients undergoing cataract surgery were implanted with a low add (+2.75 Diopters [D]) bifocal (Tecnis ZKB00; Johnson and Johnson Surgical Vision Inc., Jacksonville, Florida, USA) IOL (MIOL Group).
  Interventions: Device: Tecnis +2.75 D (ZKB00) and Tecnis Symfony (ZXR00)
- EDOF Group (Active Comparator): 30 eyes of 15 cataract patients undergoing cataract surgery were implanted with an EDOF (Tecnis Symfony [ZXR00]; Johnson and Johnson Surgical Vision Inc., Jacksonville, Florida, USA) IOL (EDOF Group).
  Interventions: Device: Tecnis +2.75 D (ZKB00) and Tecnis Symfony (ZXR00)

INTERVENTIONS:
Device: Tecnis +2.75 D (ZKB00) and Tecnis Symfony (ZXR00) — This study included 30 eyes of 15 cataract patients undergoing cataract surgery with implantation of a low add (+2.75 Diopters [D]) bifocal (Tecnis ZKB00; Johnson and Johnson Surgical Vision Inc., Jacksonville, Florida, USA) IOL (MIOL Group) and 30 eyes of 15 patients with implantation of an EDOF (Tecnis Symfony [ZXR00]; Johnson and Johnson Surgical Vision Inc., Jacksonville, Florida, USA) IOL (EDOF Group).

SUMMARY:
The innovations in phacoemulsification surgery and advances in surgical equipment ensure a safe extraction of the crystalline lens and implantation of intraocular lenses (IOL). As a result of developing intraocular lens technologies and changing patient demands, many multifocal, accommodative, toric, toric-multifocal, and extended depth of focus (EDOF) IOLs have been introduced and the original aim of restoration of far vision with implanted monocular IOLs has been evolved to an objective of improved vision at different distances with total spectacle independence. This study aimed to compare the visual acuity at different distances, contrast sensitivity, spectacle needs, photic phenomena, and quality of life parameters of patients bilaterally implanted with a low add bifocal (Tecnis ZKB00) or an EDOF IOL (Tecnis Symfony), both with planned mini-monovision to improve near vision.

DETAILED DESCRIPTION:
The innovations in phacoemulsification surgery and advances in surgical equipment ensure a safe extraction of the crystalline lens and implantation of intraocular lenses (IOL). As a result of developing intraocular lens technologies and changing patient demands, many multifocal, accommodative, toric, toric-multifocal, and extended depth of focus (EDOF) IOLs have been introduced and the original aim of restoration of far vision with implanted monocular IOLs has been evolved to an objective of improved vision at different distances with total spectacle independence. This study aimed to compare the visual acuity at different distances, contrast sensitivity, spectacle needs, photic phenomena, and quality of life parameters of patients bilaterally implanted with a low add bifocal (Tecnis ZKB00) or an EDOF IOL (Tecnis Symfony), both with planned mini-monovision to improve near vision. In this regard, binocular logMAR uncorrected visual acuities (UVA), monocular defocus curves, CS with CSV 1000-E and Pelli-Robson Test (PRT), spectacle needs and quality of life parameters with NEI RQL-42 questionnaire were evaluated at postoperative 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were patients with bilateral visually significant cataract seeking spectacle independence, especially at far and intermediate distances, age of ≥18 years, preoperative corneal astigmatism less than 1.00 D, axial length (AL) between 21 - 26.5 mm, and availability to attend all follow-up visits.

Exclusion Criteria:

Patients were excluded from the study if any of the following conditions were present: high visual demand for near vision, amblyopia, glaucoma, corneal opacity, severe/moderate to severe dry eye, pupillary abnormalities and dysfunction, corneal astigmatism ≥1.00 D, AL <21 mm or ≥26.5 mm, diabetes mellitus with retinal changes, active uveitis or history of uveitis, previous ocular surgery and lack of attendance to any follow-up visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
The visual acuity | Preoperative
  monocular and binocular uncorrected and corrected distance (UDVA, CDVA; at 6 m), intermediate (UIVA, CIVA; at 60 cm), and near (UNVA, CNVA; at 40 cm) logMAR visual acuity were assessed with electronic shelled chart.Distance visual acuity was measured with LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Snellen Charts under photopic conditions (85 cd/m2). Intermediate and near visual acuities were measured and recorded with a Turkish reading chart prepared with reference to Bailey-Lovie and ETDRS (Early Treatment Diabetic Retinopathy Study) reading charts covering international standards.13 The logMAR values of the chart designed for 35 cm distance were corrected with the formula "log10(standard distance/new distance [cm])" according to the distance used (40 and 60 cm).
The visual acuity | Postoperative 1st month
  monocular and binocular uncorrected and corrected distance (UDVA, CDVA; at 6 m), intermediate (UIVA, CIVA; at 60 cm), and near (UNVA, CNVA; at 40 cm) logMAR visual acuity were assessed with electronic shelled chart.Distance visual acuity was measured with LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Snellen Charts under photopic conditions (85 cd/m2). Intermediate and near visual acuities were measured and recorded with a Turkish reading chart prepared with reference to Bailey-Lovie and ETDRS (Early Treatment Diabetic Retinopathy Study) reading charts covering international standards.13 The logMAR values of the chart designed for 35 cm distance were corrected with the formula "log10(standard distance/new distance [cm])" according to the distance used (40 and 60 cm).
The visual acuity | Postoperative 3rd month
  monocular and binocular uncorrected and corrected distance (UDVA, CDVA; at 6 m), intermediate (UIVA, CIVA; at 60 cm), and near (UNVA, CNVA; at 40 cm) logMAR visual acuity were assessed with electronic shelled chart.Distance visual acuity was measured with LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Snellen Charts under photopic conditions (85 cd/m2). Intermediate and near visual acuities were measured and recorded with a Turkish reading chart prepared with reference to Bailey-Lovie and ETDRS (Early Treatment Diabetic Retinopathy Study) reading charts covering international standards.13 The logMAR values of the chart designed for 35 cm distance were corrected with the formula "log10(standard distance/new distance [cm])" according to the distance used (40 and 60 cm).
The visual acuity | Postoperative 6th month
  monocular and binocular uncorrected and corrected distance (UDVA, CDVA; at 6 m), intermediate (UIVA, CIVA; at 60 cm), and near (UNVA, CNVA; at 40 cm) logMAR visual acuity were assessed with electronic shelled chart.Distance visual acuity was measured with LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Snellen Charts under photopic conditions (85 cd/m2). Intermediate and near visual acuities were measured and recorded with a Turkish reading chart prepared with reference to Bailey-Lovie and ETDRS (Early Treatment Diabetic Retinopathy Study) reading charts covering international standards.13 The logMAR values of the chart designed for 35 cm distance were corrected with the formula "log10(standard distance/new distance [cm])" according to the distance used (40 and 60 cm).
The contrast sensitivity (CS), | Preoperative
  Contrast sensitivity (CS) was evaluated at 3, 6, 12 and 18 cycle per degree (cpd) spatial frequencies with CSV-1000 E test (VectorVision, Ohio, USA) under mesopic (3.5 candela [cd]/m2) conditions at 2.5 m with distance refractive correction. The test was conducted with and without glare, and as a glare source, two halogen lamps located either side of the test chart and producing 2.5 cd/m2 luminance at eye plane were used. CS at different spatial frequencies was compared with the physiologic CS range for normal subjects of similar age. CS was also evaluated with the LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Pelli-Robson Test (PRT) under photopic (85 cd/m2) and mesopic (3.5 cd/m2) conditions at 3 m monocularly with distance refractive correction. To the best of our knowledge, PRT CS normal values, performed under similar conditions, are not available in the literature, so the data was used only for intergroup comparisons.
The contrast sensitivity (CS), | Postoperative 1st month
  Contrast sensitivity (CS) was evaluated at 3, 6, 12 and 18 cycle per degree (cpd) spatial frequencies with CSV-1000 E test (VectorVision, Ohio, USA) under mesopic (3.5 candela [cd]/m2) conditions at 2.5 m with distance refractive correction. The test was conducted with and without glare, and as a glare source, two halogen lamps located either side of the test chart and producing 2.5 cd/m2 luminance at eye plane were used. CS at different spatial frequencies was compared with the physiologic CS range for normal subjects of similar age. CS was also evaluated with the LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Pelli-Robson Test (PRT) under photopic (85 cd/m2) and mesopic (3.5 cd/m2) conditions at 3 m monocularly with distance refractive correction. To the best of our knowledge, PRT CS normal values, performed under similar conditions, are not available in the literature, so the data was used only for intergroup comparisons.
The contrast sensitivity (CS), | Postoperative 3rd month
  Contrast sensitivity (CS) was evaluated at 3, 6, 12 and 18 cycle per degree (cpd) spatial frequencies with CSV-1000 E test (VectorVision, Ohio, USA) under mesopic (3.5 candela [cd]/m2) conditions at 2.5 m with distance refractive correction. The test was conducted with and without glare, and as a glare source, two halogen lamps located either side of the test chart and producing 2.5 cd/m2 luminance at eye plane were used. CS at different spatial frequencies was compared with the physiologic CS range for normal subjects of similar age. CS was also evaluated with the LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Pelli-Robson Test (PRT) under photopic (85 cd/m2) and mesopic (3.5 cd/m2) conditions at 3 m monocularly with distance refractive correction. To the best of our knowledge, PRT CS normal values, performed under similar conditions, are not available in the literature, so the data was used only for intergroup comparisons.
The contrast sensitivity (CS), | Postoperative 6th month
  Contrast sensitivity (CS) was evaluated at 3, 6, 12 and 18 cycle per degree (cpd) spatial frequencies with CSV-1000 E test (VectorVision, Ohio, USA) under mesopic (3.5 candela [cd]/m2) conditions at 2.5 m with distance refractive correction. The test was conducted with and without glare, and as a glare source, two halogen lamps located either side of the test chart and producing 2.5 cd/m2 luminance at eye plane were used. CS at different spatial frequencies was compared with the physiologic CS range for normal subjects of similar age. CS was also evaluated with the LCD screen version (CSO Vision Chart, Mod CVC02, version 1.3.0, Florence, Italy) of Pelli-Robson Test (PRT) under photopic (85 cd/m2) and mesopic (3.5 cd/m2) conditions at 3 m monocularly with distance refractive correction. To the best of our knowledge, PRT CS normal values, performed under similar conditions, are not available in the literature, so the data was used only for intergroup comparisons.
Quality of life measurement | Preoperative
  Quality of life parameters were evaluated by the validated Turkish version of the National Eye Institute Refractive Error Quality of Life Instrument 42 (NEI RQL-42) questionnaire. It includes 13 subscales of quality of life parameters calculated according to a scoring key, and a "total score" can be obtained by calculating the mean value of all 42 questions.
Quality of life measurement | Postoperative 1st month
  Quality of life parameters were evaluated by the validated Turkish version of the National Eye Institute Refractive Error Quality of Life Instrument 42 (NEI RQL-42) questionnaire. It includes 13 subscales of quality of life parameters calculated according to a scoring key, and a "total score" can be obtained by calculating the mean value of all 42 questions.
Quality of life measurement | Postoperative 3rd month
  Quality of life parameters were evaluated by the validated Turkish version of the National Eye Institute Refractive Error Quality of Life Instrument 42 (NEI RQL-42) questionnaire. It includes 13 subscales of quality of life parameters calculated according to a scoring key, and a "total score" can be obtained by calculating the mean value of all 42 questions.
Quality of life measurement | Postoperative 6th month
  Quality of life parameters were evaluated by the validated Turkish version of the National Eye Institute Refractive Error Quality of Life Instrument 42 (NEI RQL-42) questionnaire. It includes 13 subscales of quality of life parameters calculated according to a scoring key, and a "total score" can be obtained by calculating the mean value of all 42 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ebru Toker, Professor, Study Director — Marmara University
Locations (1):
- Marmara University School of Medicine, Department of Ophthalmology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Rosen E, Alio JL, Dick HB, Dell S, Slade S. Efficacy and safety of multifocal intraocular lenses following cataract and refractive lens exchange: Metaanalysis of peer-reviewed publications. J Cataract Refract Surg. 2016 Feb;42(2):310-28. doi: 10.1016/j.jcrs.2016.01.014. PMID 27026457
- [Background] Kim JS, Jung JW, Lee JM, Seo KY, Kim EK, Kim TI. Clinical Outcomes Following Implantation of Diffractive Multifocal Intraocular Lenses With Varying Add Powers. Am J Ophthalmol. 2015 Oct;160(4):702-9.e1. doi: 10.1016/j.ajo.2015.07.021. Epub 2015 Jul 21. PMID 26209232
- [Background] Kretz FT, Gerl M, Gerl R, Muller M, Auffarth GU; ZKB00 Study Group. Clinical evaluation of a new pupil independent diffractive multifocal intraocular lens with a +2.75 D near addition: a European multicentre study. Br J Ophthalmol. 2015 Dec;99(12):1655-9. doi: 10.1136/bjophthalmol-2015-306811. Epub 2015 May 18. PMID 25987651
- [Background] Pedrotti E, Bruni E, Bonacci E, Badalamenti R, Mastropasqua R, Marchini G. Comparative Analysis of the Clinical Outcomes With a Monofocal and an Extended Range of Vision Intraocular Lens. J Refract Surg. 2016 Jul 1;32(7):436-42. doi: 10.3928/1081597X-20160428-06. PMID 27400074